CLINICAL TRIAL: NCT06179069
Title: An Open-label, Multicenter Study of ZL-1310 to Evaluate the Safety, Efficacy, and Pharmacokinetics in Participants With Small Cell Lung Cancer
Brief Title: A Study of ZL-1310 in Subjects With Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Collaborators: Zai Lab (US) LLC (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1310-001
Record Dates: First submitted 2023-12-07; First posted 2023-12-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: SCLC
MeSH Terms: interventions — atezolizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (10):
- Dose Escalation: Part 1A (Experimental): ZL-1310 as a single-agent
  Interventions: Drug: ZL-1310
- Dose Expansion: Part 1B (Experimental): ZL-1310 in combination with Atezolizumab
  Interventions: Drug: ZL-1310; Drug: Atezolizumab
- Dose Escalation: Part 1C (Experimental): ZL-1310 in combination with Atezolizumab and Carboplatin as induction and followed by ZL-1310 and Atezolizumab as maintenance
  Interventions: Drug: ZL-1310; Drug: Atezolizumab; Drug: Carboplatin
- Dose Expansion: Arm 1 (Part 2) (Experimental): Dose level 1 of ZL-1310 established from single-agent dose-escalation
  Interventions: Drug: ZL-1310
- Dose Expansion: Arm 2 (Part 2) (Experimental): Dose level 2 of ZL-1310 established from single-agent dose escalation
  Interventions: Drug: ZL-1310
- Dose Extension: Arm 1 (Part 2) (Experimental): ZL-1310 as a single agent
  Interventions: Drug: ZL-1310
- Doublet Dose Optimization: Arm 1 (Part 3) (Experimental): Dose level 1 of ZL-1310 established from single agent dose escalation, in combination with Atezolizumab
  Interventions: Drug: ZL-1310; Drug: Atezolizumab
- Doublet Dose Optimization: Arm 2 (Part 3) (Experimental): Dose level 2 of ZL-1310 established from single agent dose escalation in combination with Atezolizumab
  Interventions: Drug: ZL-1310; Drug: Atezolizumab
- Triplet Dose Optimization: Arm 1 (Part 4) (Experimental): Dose level 1 of ZL-1310 established from single agent dose escalation in combination with Atezolizumab + Carboplatin induction followed by ZL-1310 + Atezolizumab as maintenance
  Interventions: Drug: ZL-1310; Drug: Atezolizumab; Drug: Carboplatin
- Triplet Dose Optimization: Arm 2 (Part 4) (Experimental): Dose level 2 of ZL-1310 established from single agent dose escalation, in combination with Atezolizumab + Carboplatin induction followed by ZL-1310 + atezolizumab as induction
  Interventions: Drug: ZL-1310; Drug: Atezolizumab; Drug: Carboplatin

INTERVENTIONS:
Drug: ZL-1310 — Drug: ZL-1310
Drug: Atezolizumab — Drug Atezolizumab
  Arms: Dose Escalation: Part 1C; Dose Expansion: Part 1B; Doublet Dose Optimization: Arm 1 (Part 3); Doublet Dose Optimization: Arm 2 (Part 3); Triplet Dose Optimization: Arm 1 (Part 4); Triplet Dose Optimization: Arm 2 (Part 4)
Drug: Carboplatin — Drug Carboplatin
  Arms: Dose Escalation: Part 1C; Triplet Dose Optimization: Arm 1 (Part 4); Triplet Dose Optimization: Arm 2 (Part 4)

SUMMARY:
An open-label, multicenter study of ZL-1310 as a single agent and in combination with Atezolizumab (with and without Carboplatin) to evaluate the safety, efficacy, and pharmacokinetics in subjects with small cell lung cancer

DETAILED DESCRIPTION:
This is an open-label, ascending, multiple-dose, phase 1 study evaluating ZL-1310 as a single agent, in combination with Atezolizumab, and in combination with Atezolizumab and Carboplatin in subjects with extensive SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Participant with metastatic or extensive-stage small cell lung cancer (de novo, not transformed) and for Part 1A and 1B must have documented disease progression during or following a platinum-based chemotherapy regimen. For Part 1C and Part 4, no prior systemic treatment for SCLC (including chemoradiotherapy for limited-stage SCLC). For Part 1B backfill, first-line setting: no prior systemic treatment for SCLC (including chemoradiotherapy for limited-stage SCLC); or, first-line maintenance setting: participants have received at least 4 cycles of 1L induction therapy with carboplatin or cisplatin, etoposide, and anti-PD-L1 inhibitor for ES-SCLC with ongoing CR, PR, or SD per RECIST v1.1 assessed by the investigator. For Part 3, participants have received at least 4 cycles of 1L induction therapy with carboplatin or cisplatin etoposide, and anti-PD-L1 inhibitor for ES-SCLC with ongoing CR, PR, or SD per RECIST v1.1 assessed by the investigator.
* Adult men and women ≥18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Subjects must have at least one measurable target lesion as defined by RECIST v1.1 on CT, PET/CT, or MRI.
* Subjects must be willing to undergo a tumor biopsy or must provide archived tumor tissue sample at screening per protocol guidelines.
* Life Expectancy >/= 3 months.

Exclusion Criteria:

* Participants with another known malignancy that is progressing or requires active treatment within the last 2 years. Exceptions: basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin with previously administered curative treatment, in situ cervical cancer, or other cancers that do not require systemic anti-cancer therapies and will not impact life expectancy.
* Symptomatic or untreated brain metastasis requiring concurrent treatment. For Part 2, Part 3, and Part 4 the following subjects can be enrolled if they have a stable neurologic status for at least 2 weeks prior to the first dose of ZL-1310:

  1. Subjects with untreated and asymptomatic brain metastases.
  2. Subjects with treated brain metastases that are no longer symptomatic (i.e. without neurologic signs or symptoms), who require no treatment with steriods or anticonvulsants and have recovered from the actue toxic effects of radiotherapy.
* Subjects with leptomeningeal disease.
* Treatment with any systemic anti-cancer treatment or other investigational products/ device within 3 weeks before first dose of study treatment.
* Non-palliative radiotherapy within 2 weeks prior to first dose of study treatment or have had a history of radiation pneumonitis.
* Major surgery within 4 weeks of the first dose of study treatment.
* Hypersensitivity to any ingredient of the study treatment.
* Inadequate organ function (as defined in protocol) within 10 days prior to the first dose of study treatment,
* Participants with a diagnosis of immunodeficiency or receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 14 days or 5 half-lives before the first dose of study treatment, whichever is longer.
* Participants have received a live or live-attenuated vaccine within 30 days of planned start of study therapy.
* Impaired cardiac function or clinically significant cardiac disease within the last 3 months before administration of the first dose of the study treatment
* Lung-specific intercurrent clinically significant illnesses and any autoimmune, connective tissue, or inflammatory disorders, including but not limited to pneumonitis.
* Pregnant or nursing (lactating) women.
* Participants who have been on concomitant strong CYP3A or CYP2D6 inhibitors within 14 days or 5 half-lives before the first study treatment, whichever is longer.
* For Part 1C and Part 4 (ZL-1310 in combination with Atezolizumab and Carboplatin), participants who received prior treatment with CD137 agonists or immune checkpoint blockade therapies, anti-PD-1, and anti-PD-L1 therapeutic antibodies.
* For Part 1B (ZL-1310 in combination with Atezolizumab) and Part 1C (ZL-1310 in combination with Atezolizumab and Carboplatin), participants who received systemic immunostimulatory agents (including but not limited to, IFNs and IL2) within 4 weeks or 5 drug-elimination half-lives, whichever is longer, prior to the initiation of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2027-05-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities of ZL-1310 as a single agent (Part 1A), in combination with Atezolizumab (Part 1B), and in combination with atezolizumab and carboplatin (Part 1C) | up to 24 months
  Number of subjects with Dose Limiting Toxicities (DLTs)
Incidence of Treatment Emergent Adverse-Events of ZL-1310 as a single agent (Part 1A), in combination with atezolizumab (Part 1B), and in combination with atezolizumab and carboplatin (Part 1C) | up to 24 months
  Number of subjects with treatment-emergent adverse events (TEAEs)
Incidence of Serious Adverse Events of ZL-1310 as a single agent (Part 1A), in combination with atezolizumab (Part 1B), and in combination with atezolizumab and carboplatin (Part 1C) | up to 24 months
  Number of subjects with serious adverse events
Incidence of Treatment Emergent Adverse Events of ZL-1310 as a single agent (Part 2), in combination with atezolizumab (Part 3) and in combination with atezolizumab and carboplatin (Part 4) | up to 24 months
  Number of subjects with treatment emergent adverse events leading to dose modifications and/or study treatment discontinuation
Incidence of Serious Adverse-Events (SAEs) of ZL-1310 as a single agent (Part 2), in combination with atezolizumab (Part 3), and in combination with atezolizumab and carboplatin (Part 4) | up to 24 months
  Number of subjects with serious adverse events
Antitumor activity per RECIST v1.1 by investigator's assessment of ZL-1310 as a single agent (Part 2), in combination with atezolizumab (Part 3), and in combination with atezolizumab and carboplatin (Part 4) | up to 24 months
  antitumor activity per RECIST v1.1 by investigator's assessment
Objective response rate (ORR) per RECIST v1.1 of ZL-1310 as a single agent (Part 2) and in combination with atezolizumab and carboplatin (Part 4) | up to 24 months
  objective response rate per RECIST v1.1
Disease control rate (DCR) per RECIST v1.1 of ZL-1310 in combination with atezolizumab | up to 24 months
  disease control rate per RECIST v1.1

SECONDARY OUTCOMES:
Objective response rate (ORR) per RECIST 1.1 of ZL-1310 as a single agent (Part 1A) in combination with atezolizumab (Part 1B), in combination with atezolizumab and carboplatin (Part 1C, Part 3) | up to 24 months
  Objective Response Rate (ORR) per RECIST 1.1
Disease control rate (DCR) per RECIST v1.1 of ZL-1310 as a single agent (Part 1A and Part 2), in combination with atezolizumab (Part 1B), and in combination with atezolizumab and carboplatin (Part 4) | up to 24 months
  Disease control rate (DCR) per RECIST v1.1
Duration of response per RECIST v1.1 | up to 24 months
  Duration of response per RECIST v1.1
Progression free survival per RECIST v1.1 | up to 24 months
  Progression free survival per RECIST v1.1
Overall Survival of ZL-1310 | up to 24 months
  Overall Survival of ZL-1310
Pharmacokinetics: Total Antibody of ZL-1310 | up to 24 months
  Pharmacokinetics: Total Antibody of ZL-1310
Pharmacokinetics: Unconjugated payloads of ZL-1310 | up to 24 months
  Pharmacokinetics: Unconjugated payloads of ZL-1310

CONTACTS AND LOCATIONS:
Locations (38):
- United States (11):
  - Zai Lab Site 2005, Duarte, California
  - Zai Lab Site 2030, New Haven, Connecticut
  - Zai Lab Site 2026, Sarasota, Florida
  - Zai Lab Site 2013, Detroit, Michigan
  - Zai Lab Site 2001, Hackensack, New Jersey
  - Zai Lab Site 2002, Buffalo, New York
  - Zai Lab Site 2018, Durham, North Carolina
  - Zai Lab Site 2024, Cleveland, Ohio
  - Zai Lab Site 2029, Pittsburgh, Pennsylvania
  - Zai Lab Site 2012, Charleston, South Carolina
  - Zai Lab Site 2006, Fairfax, Virginia
- China (16):
  - Zai Lab Site 1004, Hefei, Anhui
  - Zai Lab Site 1005, Beijing, Beijing Municipality
  - Zai Lab Site 1012, Xiamen, Fujian
  - Zai Lab Site 1001, Guangzhou, Guangdong
  - Zai Lab Site 1009, Harbin, Heilongjiang
  - Zai Lab Site 1006, Zhengzhou, Henan
  - Zai Lab 1002, Wuhan, Hubei
  - Zai Lab Site 1014, Changsha, Hunan
  - Zai Lab Site 1016, Nanjing, Jiangsu
  - Zai Lab Site 1003, Nanchang, Jiangxi
  - Zai Lab Site 1008, Ch’ang-ch’un, Jilin
  - Zai Lab Site 1017, Shenyang, Liaoning
  - Zai Lab Site 1015, Xi'an, Shaanxi
  - Zai Lab Site 1011, Jinan, Shandong
  - Zai Lab Site 1010, Shanghai, Shanghai Municipality
  - Zai Lab Site 1013, Chengdu, Sichaun
- Spain (11):
  - Zai Lab Site 8002, Barcelona, Barcelona
  - Zai Lab Site 8003, Madrid, Madrid
  - Zai Lab Site 8006, Madrid, Madrid
  - Zai Lab Site 8005, Seville, Sevilla
  - Zai Lab Site 8004, Valencia, Valencia
  - Zai Lab Site 8001, Valencia, Valencia
  - Zai Lab Site 8007, Barcelona
  - Zai Lab Site 8009, Madrid
  - Zai Lab Site 8008, Málaga
  - Zai Lab Site 8010, Pozuelo de Alarcón
  - Zai Lab Site 8011, Seville

IPD SHARING:
Plan to Share IPD: No